CLINICAL TRIAL: NCT03429803
Title: A Phase I Study of Tovorafenib/DAY101 (Formerly TAK-580, MLN2480) for Children With Low-Grade Gliomas and Other RAS/RAF/MEK/ERK Pathway Activated Tumors
Brief Title: DAY101 In Gliomas and Other Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karen D. Wright, MD (Other)
Collaborators: PLGA Fund at Pediatric Brain Tumor Foundation (Unknown); National Cancer Institute (NCI) (NIH); Pacific Pediatric Neuro-Oncology Consortium (Other); Team Jack Foundation (Unknown); Day One Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Karen D. Wright, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-589; P50CA165962 (NIH); PNOC014 (Other: Pacific Pediatric Neuro-Oncology Consortium)
Record Dates: First submitted 2018-01-09; First posted 2018-02-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Low-grade Glioma
Keywords: low-grade glioma
MeSH Terms: interventions — tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DAY101 (formerly TAK-580, MLN2480) BSA </= 1.5m^2 (Experimental): Phase I Part B BSA </= 1.5m^2
  * Patients (< 25 years) with radiographically recurrent or radiographically progressive non-hematologic malignancies (Central Nervous System (CNS) or solid tumors) associated with activation of the RAS/RAF/MEK/ERK pathway will be eligible with the exception of patients with NF1
  * Study treatment cycle lasts 28 days, oral, once a week
  Interventions: Drug: DAY101
- DAY101 (formerly TAK-580, MLN2480) BSA > 1.5m^2 (Experimental): Phase I Part B BSA > 1.5m^2
  * Patients (< 25 years) with radiographically recurrent or radiographically progressive non-hematologic malignancies (Central Nervous System (CNS) or solid tumors) associated with activation of the RAS/RAF/MEK/ERK pathway will be eligible with the exception of patients with NF1
  * Study treatment cycle lasts 28 days, oral, once a week
  Interventions: Drug: DAY101

INTERVENTIONS:
Drug: DAY101 — 28 day cycle, oral, once per week
  Other Names: MLN2480; TAK-580

SUMMARY:
This research study is studying a drug Tovorafenib/DAY101 (formerly TAK-580, MLN2480) as a possible treatment a low-grade glioma that has not responded to other treatments.

The name of the study drug involved in this study is:

• Tovorafenib/DAY101 (formerly TAK-580, MLN2480)

DETAILED DESCRIPTION:
This is a Phase I clinical trial. A Phase I clinical trial tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved DAY101 as a treatment for any disease.

This is the first time that DAY101 will be given to children. There is limited experience with DAY101 in humans.

The purpose of this study is to test the safety DAY101 in children and adolescent participants with brain tumors. The investigators want to find out what effects, good and/or bad, it has on participants and the participant's brain tumor, and find the dose of DAY101 that is tolerated by participants without too many side effects to use in Phase II of the study.

Research in the laboratory has shown that DAY101 may have activity against cancer cells. DAY101 belongs to a group of drugs called type II BRAF inhibitors. BRAF abnormalities are found in cancer cells. There are no type II BRAF inhibitors approved by the FDA for humans at the time of this study's start. DAY101 functions by binding the mutant BRAF molecule and causing a conformation change in the molecule thereby blocking the signal that tells the tumor cell to divide.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:

  * Phase I

    * Pediatric patients with radiographically recurrent or radiographically progressive non-hematologic malignancies (Central Nervous System (CNS) or solid tumors) associated with activation of the RAS/RAF/MEK/ERK pathway will be eligible with the exception of patients with NF1.
    * Mutational status requires a pathology report, genomic sequencing, or immunohistochemical report of a mutation or activation of the RAS/RAF/MEK/ERK pathway.
  * The remaining criteria include:

    * Patients must be >1 year and <25 years old.
    * Patients must have adequate performance status:

      * Karnofsky ≥ 50 for patients ≥ 16 years of age (See Appendix A).
      * Lansky ≥ 50 for patients < 16 years of age (See Appendix A).
    * Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score (See Appendix A).
    * A patient who has failed standard therapy. Note: standard of care for resectable low grade glioma, as an example, is surgery. Therefore, patients with low grade glioma that recurs after presumed gross total resection may enroll without prior chemotherapy exposure.
    * At least 1 measurable lesion that can be reproducibly measured in 2 dimensions
    * Previous chemotherapy and hormone therapy (excluding physiologic replacement) must be completed at least 4 weeks or 4 half-lives, whichever is longer, prior to administration of DAY101.
    * Previous immunotherapy/ monoclonal antibody use must be completed at least 4 weeks or 4 half lives, whichever is longer prior to administration of DAY101.
    * Previous MEK or BRAF inhibitors must be completed at least 7 days prior to the administration of DAY101.
    * Focal or cranial spinal irradiation to the target lesion (whether as treatment or palliation) must be completed at least 6 months prior to administration of DAY101 to address the possibility of pseudoprogression. If pseudoprogression is definitively ruled out with tissue sampling (biopsy or repeat surgery), the patient may enroll after completion of radiation therapy at time of defined progression (and not wait 6 months) as long as patient meets other eligibility requirements.
    * All associated toxicities from previous therapies must be resolved to ≤ Grade 1 or considered baseline prior to administration of DAY101.
    * Female patients who:

      * Are postmenopausal for at least 1 year before the screening visit, OR
      * Are surgically sterile, OR
      * If they are of childbearing potential, agree to practice 1 effective method of contraception and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer as mandated by local labeling [e.g., United States Protection and Investigations (USPI), Summary of Product Characteristics (SmPC), etc,]) after the last dose of study drug, OR
      * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
    * Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

      * Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
      * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
      * Agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
    * Patient must be able to swallow pills whole.
    * Patient, parent, or legal guardian must be able to understand and be willing to provide informed consent.
    * Thyroid function tests must be consistent with stable thyroid function. Patients on a stable dose of thyroid replacement therapy for a suggested minimum of 3 weeks before Cycle 1, Day 1 are eligible.
    * Left ventricular ejection fraction (LVEF) of 50% or greater, as measured by echocardiogram (ECHO) or multiple gated acquisition (MUGA) scan, within 28 days before the first dose of DAY101
    * Inclusion of Women, Minorities, and Other Underrepresented Populations: This protocol is open to males and females of all races. See inclusion criteria above regarding specific eligibility requirements for female and male patients of child-bearing or child-fathering potential, respectively.
* Exclusion Criteria: Patients with any of the following characteristics will NOT be eligible:

  * Patients with clinical progression but without radiographically recurrent or radiographically progressive disease.
  * Patients with NF1
  * History of any major disease that might interfere with safe protocol participation, as determined by the investigator
  * Patients with a history or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO), or ophthalmopathy present at baseline that would be considered a risk factor for CSR or RVO

    --- Patients with history of Drug Rash with Eosinophilia and Systemic Symptoms (DRESS) or Steven Johnson Syndrome in the setting of prior MEK or BRAF inhibitor exposure
  * Laboratory values:

    * Absolute neutrophil count (ANC) ≤ 1000/μL
    * Platelet count ≤ 75,000/μL (transfusion independent)
    * Hemoglobin < 9 g/dL (hemoglobin may be supported by transfusion, erythropoietin, or other approved hematopoietic growth factors)
    * Serum bilirubin ≥ 1.5 × upper limit of normal (ULN) or ³ 2 ´ ULN if patient is known to have Gilbert's Disease as the only underlying hepatic disorder
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.5 × ULN. AST and ALT ≥ 5 × ULN for patients with liver metastasis
    * Serum creatinine ≥ 2.0 mg/dL
  * Current enrollment in any other investigational treatment study
  * Evidence of current uncontrolled cardiovascular conditions, including but not limited to clinically significant cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction, within the past 6 months
  * Active hepatitis or human immunodeficiency virus infection
  * Active bacterial or viral infection
  * Female patients who are pregnant or currently breastfeeding. Female patients of childbearing potential must have a negative serum pregnancy test prior to enrollment.
  * Major surgery within 28 days of Day 1 (does not include central venous access or shunts)
  * Inability to comply with study requirements
  * Refractory nausea and vomiting, malabsorption, or significant bowel or stomach resection that would preclude adequate absorption of DAY101
  * Treatment with any of the strong CYP2C inducers within 14 days before the first dose of DAY101 (see Appendix H).
  * Treatment with gemfibrozil (strong CYP2C8 inhibitor) within 14 days before the first dose of DAY101.
  * Other unspecified reasons that, in the opinion of the investigator, make the patient unsuitable for enrollment.
  * Important note: The eligibility criteria listed above are interpreted literally and cannot be waived.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Greater and equal 28 days
  A DLT is defined as an AE assessed as at least possibly related to the study medication, which occurs during Cycle 1 (typically 28 days following the first dose of DAY101)

SECONDARY OUTCOMES:
Blood samples for DAY101 concentration measurements (i.e. pharmacokinetic measures) | cycle 1 day 1 1-4 hours post dose; cycle 1 day 3-6 random level; cycle 2 day 1 pre-dose; cycle 3 day 1 random level; end of therapy or at time of toxicity requiring patient be taken off study or dose held; time of surgery if applicable)
  measurement of phosphorylated ERK in peripheral blood mononuclear cells, will be performed on all patients in the phase I component of the trial
Best Overall Response | 48 Weeks
  Pediatric patients (>1 year and <25 years of age). each evaluable patient will be classified as either a responder (complete response, partial response, or stable disease) or a non-responder (<stable disease)
Number of participants with adverse events | 48 Weeks
  Frequency of adverse events (AEs) with once weekly administration of DAY101
Number of participants with serious adverse events | 48 weeks
  Frequency of serious adverse events (SAEs) with once weekly administration of DAY101

CONTACTS AND LOCATIONS:
Overall Officials: Karen D. Wright, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (15):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massacusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institite, Boston, Massachusetts
  - Children's Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
o The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu